CLINICAL TRIAL: NCT00251342
Title: Outcome of Postnatal Depression Screening Using Edinburgh Postnatal Depression Scale
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Hong Kong Department of Health (Unknown); The University of Hong Kong (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: CRE-2005.224-T; CUHK_CCT00019
Record Dates: First submitted 2005-11-09; First posted 2005-11-10 (Estimated); Last update posted 2007-04-05 (Estimated); Status verified 2007-04

CONDITIONS: Depression, Postpartum
Keywords: Postnatal depression; Randomized controlled trial; Screening; Outcome; Edinburgh Postnatal Depression Scale
MeSH Terms: conditions — Depression, Postpartum | interventions — Psychiatric Status Rating Scales

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Edinburgh Postnatal Depression Scale

SUMMARY:
The objective of the present study is to evaluate the effectiveness of postnatal depression screening by comparing the mental health outcome (at 6 months postpartum) of mothers under the Edinburgh Postnatal Depression Scale (EPDS) screening programme versus usual clinical practice (usual practice), using randomized controlled trial design. With the use of the EPDS for the screening of postnatal depression, it is expected that more mothers in need of intervention (including mental health intervention, guidance in childcare and parenting, counseling in family relationships, etc) will be picked up and offered appropriate intervention, compared to the usual practice. It is hypothesized that the mental health of the group of women under the EPDS screening programme will be better than those under the usual practice, on subsequent follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese mothers of newborn babies <= 2 months who are registered with the 4 Maternal and Child Health Centres under study;
2. Normally resident in Hong Kong (Hong Kong ID card holder, or HK Birth Certificate [with status of permanent resident indicated established] holder, or people who have been granted unconditional stay in Hong Kong, or passport holders having valid travel document showing the right to land in Hong Kong, or permission to land, or eligibility of HK permanent ID card verified, or entitlement to the right of abode in HK)

Exclusion Criteria:

1. Those who do not use the Chinese language (in both the written and spoken form);
2. Those who are under active psychiatric contact;
3. Those who delivered in hospitals which are still conducting their own EPDS screening programme.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 460
Dates: Start 2005-10; Study Completion 2008-01 (Estimated)

PRIMARY OUTCOMES:
Mother's mental health at 6 months postpartum, as measured on the EPDS and General Health Questionnaire-12 (GHQ-12), both being self-report questionnaires.

SECONDARY OUTCOMES:
Mother's parenting stress (measured by the Parenting Stress Index, a self-report questionnaire)
Marital relationship satisfaction (measured by the Chinese Kansas Marital Satisfaction Scale, a self-report questionnaire)
Marital status and employment status (both father and mother, where applicable) at 6 and 18 months postpartum
Child health measures, including weight at 6 and 18 months, number of hospitalizations and visits to doctors within the first 6 and 18 months as reported by mother
Mother's mental health outcome (EPDS and GHQ scores) at 18 months postpartum

CONTACTS AND LOCATIONS:
Overall Officials: Dominic TS Lee, M.D., Principal Investigator — Department of Psychiatry, The Chinese University of Hong Kong; Shirley SL Leung, MPH, Principal Investigator — Family Health Service, Department of Health, HKSAR
Locations (1):
- Maternal and Child Health Centres, Department of Health, Hong Kong, China

REFERENCES:
- [Derived] Leung SS, Leung C, Lam TH, Hung SF, Chan R, Yeung T, Miao M, Cheng S, Leung SH, Lau A, Lee DT. Outcome of a postnatal depression screening programme using the Edinburgh Postnatal Depression Scale: a randomized controlled trial. J Public Health (Oxf). 2011 Jun;33(2):292-301. doi: 10.1093/pubmed/fdq075. Epub 2010 Sep 29. PMID 20884642